CLINICAL TRIAL: NCT00859092
Title: Promotion of Thickened Feeds to Manage Newborns With Feeding Difficulties
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Oelberg, M.D. (Other)
Responsible Party: Sponsor-Investigator, David Oelberg, M.D., Principal Investigator, Eastern Virginia Medical School
Organization: Eastern Virginia Medical School (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-12-FB-0305
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Swallowing Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thickening of feeds (Experimental)
  Interventions: Dietary Supplement: Simply Thick
- Removal of thickener (No Intervention)

INTERVENTIONS:
Dietary Supplement: Simply Thick — Simply Thick® added to each bottle of formula or beast milk to create nectar or honey consistency
  Other Names: Simply Thick®
  Arms: Thickening of feeds

SUMMARY:
Swallowing dysfunction and delay of oral feeding skills in premature infants significantly delay discharge from the hospital. Thickening oral formula or breast milk feeds with commercial thickeners and rice cereal has been used in some nurseries with the goal of promoting development of adequate feeding skills. The objective of this pilot study is to examine the effect of thickened feeds on premature infants with oral feeding difficulties due to dysfunction secondary to immature swallowing.

Hypotheses:

* Thickened feeds will lead to a reduction in symptoms secondary to immature swallowing in 32-40 weeks gestational age infants when compared to non-thickened feeds
* Thickened feeds will promote transition to hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. apneas and bradycardias with oral feedings
2. oxygen desaturations with oral feedings
3. excessive coughing or gagging with oral feedings

Exclusion Criteria:

1. less than 32 weeks adjusted gestational age
2. greater than 40 weeks adjusted gestational age

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Elimination of symptoms associated with immature swallowing | 2 days

SECONDARY OUTCOMES:
Promotes transition to discharge from hospital | one week

CONTACTS AND LOCATIONS:
Overall Officials: David Oelberg, MD, Principal Investigator — Children's Hospital of The King's Daughters
Locations (1):
- Sentara Norfolk General Hospital, Norfolk, Virginia, United States